CLINICAL TRIAL: NCT01894997
Title: A Comparison of the Effects of Neuromuscular Electrical Stimulation and Intermittent Pneumatic Compression on Lower Limb Haemodynamics
Brief Title: A Comparison of the Effects of Neuromuscular Electrical Stimulation and Intermittent Pneumatic Compression on Blood Flow in the Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Irish Research Council (Other); Galway Clinic (Network)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EE-NMES-DVT-334
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Venous Thrombosis
Keywords: Deep Vein Thrombosis; Neuromuscular Electrical Stimulation; Intermittent Pneumatic Compression; Doppler Ultrasound
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVT Prophylaxis (Experimental): Neuromuscular electrical stimulation is to be applied using a custom-built, two-channel stimulator (Bioelectronics Research Cluster, National University of Ireland, Galway) with a frequency of 36 Hz, a balanced biphasic waveform with a pulse width of 350μs, a ramp up time of 500ms, a contraction time of 1s and a ramp down time of 500ms. Stimulation is to be applied every 20 seconds over a period of 5 minutes.
  Intermittent pneumatic compression is to be applied using the Novamedix A-V Impulse System Model 6000 (Novamedix distribution Limited, England), programmed to deliver compression every 20 seconds at a pressure of 130 mmHg for a 3 second duration over a period of 5 minutes.
  Interventions: Device: Neuromuscular electrical stimulator; Device: AV Impulse System Model 6000

INTERVENTIONS:
Device: Neuromuscular electrical stimulator
Device: AV Impulse System Model 6000
  Other Names: Intermittent Pneumatic Compression Device

SUMMARY:
Deep Vein Thrombosis (DVT) is a life threatening condition and a serious concern among hospitalized patients, with death occurring in approximately 6% of cases. It involves the formation of a clot where stagnant blood flow occurs, predominantly in the deep veins of the legs. Three mechanisms underlie DVT, venous stasis (slowing or stopping of the blood), hypercoagulability (increased clotting) and damage to blood vessel endothelium (damage to blood vessel wall), collectively known as Virchow's triad.

Intermittent pneumatic compression (IPC) and neuromuscular electrical stimulation (NMES) have been shown to improve lower limb blood flow. However, few studies have directly compared the two methods and those that have, have used dated NMES techniques.

The objective of this study is to compare the two methods in terms of blood flow, in both a young and an older population.

DETAILED DESCRIPTION:
Deep Vein Thrombosis (DVT) is a life threatening condition and a serious concern among hospitalized patients, with death occurring in approximately 6% of cases. It involves the formation of a clot where stagnant blood flow occurs, predominantly in the deep veins of the legs. Three mechanisms underlie DVT, venous stasis (slowing or stopping of the blood), hypercoagulability (increased clotting) and damage to blood vessel endothelium (damage to blood vessel wall), collectively known as Virchow's triad.

Intermittent Pneumatic Compression (IPC) involves the use of an inflatable cuff placed around the limb. This cuff inflates and deflates intermittently in order to squeeze blood from the underlying veins. Neuromuscular Electrical Stimulation (NMES) leads to a contraction of muscles by delivering a series of controlled electrical pulses via skin surface electrodes placed over the motor points of the targeted muscle.

ELIGIBILITY:
Inclusion Criteria:

* Free from any known illness
* Between 18 and 40 years of age
* Between 55 and 65 years of age

Exclusion Criteria:

* History of heart/respiratory problems
* Pregnancy
* Presence of implants, including cardiac pacemakers and orthopaedic implants
* History of neurological disorder
* History of severe arterial disease or known dermatological problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Blood flow measurements from the lower limb | Two hours (plus or minus half an hour)
  Doppler measurements will be taken for each of the interventions.The measurement site of interest is the popliteal vein, located at the back of the knee. Peak venous velocity, time averaged mean velocity, vein cross-sectional area and volume flow will be recorded. 3 measurements of each will be taken per intervention. No measurements will be taken within the first minute of the intervention.

SECONDARY OUTCOMES:
Blood pressure | Two hours (plus or minus half an hour)
  Blood pressure will be measured throughout the study using an OMRON RX3 Plus digital automatic blood pressure monitor.
Heart rate | Two hours (plus or minus half an hour)
  Heart rate will be measured throughout the study using an OMRON RX3 Plus digital automatic blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Gearoid OLaighin, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- National University of Ireland, Galway, Galway, Ireland